CLINICAL TRIAL: NCT03167775
Title: Clinical Trial of Elemene Injection/Elemene Oral Emulusion in Combination With the Best Supportive Treatment in the Treatment of Advanced Primary Liver Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: BeiJing Yijiayi Medicine Techonoloy Co., Ltd. (Industry)
Collaborators: Dalian Holley Kingkong Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 81YY-ZLLL-16-19
Record Dates: First submitted 2017-05-22; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Advanced Primary Liver Cancer
MeSH Terms: interventions — elemene

STUDY DESIGN:
Intervention Model Description: the patients will be treated with the Elemene Injection/Elemene Oral Emulusion in Combination with the best supportive treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Elemene + the best supportive treatment (Experimental): the patients will be treated with the Elemene Injection/Elemene Oral Emulusion in Combination with the best supportive treatment .
  Interventions: Drug: Elemene Injection/Elemene Oral Emulusion

INTERVENTIONS:
Drug: Elemene Injection/Elemene Oral Emulusion

SUMMARY:
Clinical Trial of Elemene Injection/Elemene Oral Emulusion in Combination With the Best Supportive Treatment in the Treatment of Advanced Primary Liver Cancer

DETAILED DESCRIPTION:
Patients with advanced primary liver cancer will be enrolled in the trial , then the patients will be treated with the Elemene Injection/Elemene Oral Emulusion in Combination with the best supportive treatment .The purpose of the study is to evaluate the effect and safety of the Elemene Injection/Elemene Oral Emulusion in Combination with the best supportive treatment in the treatment of advanced primary liver cancer

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old，No limit on gender
* Patients who are confirmed Locally advanced or metastatic primary liver cancerin accordance with the clinical diagnostic criteria , or by pathological histology or cytology examination, Patients who are unable to accept surgery,radiofrequency ablation、TACE and local therapy ，orLocal treatment progress failed
* have systematic treatment before( including systematic chemotherapy and/or molecular targeted therapy) , but the treatment was unsuccessed and the tumor progress
* According to RECIST V1.1，1at least has one measurable lesions
* ECOG Score ≤2
* Patients who have primary liver cancer with Child - Pugh liver function grade rating A or better B(score<=7)
* Laboratory inspection basically meets the following requirements： Blood test：a. Hb>=90g/L(without blood transfusion within 14 days), b. ANC>=1.5×10^9/L, c. PLT>=60×10^9/L. Biochemical test：a. ALB>=29g/L(without blood transfusion within 14 days), b. ALT and AST <=5ULN, c. TBIL<=2ULN, d. Cr<=1.5ULN. Blood Coagulation function:PT<=ULN+6seconds.
* Life expectancy of at least 3 months
* Subjects join the study voluntarily, sign a consent form, have good compliance, and comply with follow-up.

Exclusion Criteria:

* Patients have other anti-cancer treatment ， including α-IFN，Arsenious Acid Injection and other Traditional Chinese Medicine Patent Prescription for treating cancer
* In the past or at the same time,patients were diagnosed with other malignant tumor which have not been cured. As for skin basal cell carcinoma and cervical carcinoma in situ,they can be excepted
* Patients with severe acute infection and cann't be controled , Chronic suppurative infection , body temperature>=39℃ ， Pleural effusion（medium and large） combined with infection
* Women who is pregnant or during breast feeding and not willing to contraception during the test
* Coagulation dysfunction(PT>16 seconds ， APTT>43 seconds , TT>21 seconds , Fib<2g/L) , With bleeding tendency or the presence of vital organ thrombosis (lung, brain) is receiving thrombolytic or anticoagulant therapy
* With a mental illness, or has a history of drugs abuse
* Patients accepted any experimental drugs in the past 4 weeks
* Other reasons the researchers think not suitable

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-11-28 (Actual); Primary Completion 2019-05-27 (Estimated); Study Completion 2019-11-27 (Estimated)

PRIMARY OUTCOMES:
DCR and/or 6-months survival rate | 6 months
  Disease control rate.The proportion of patients who had a best response rating of complete response, partial response, or stable disease/

SECONDARY OUTCOMES:
ORR | 1year
  Objective response rate.The proportion of patients who had a best response rating of complete response and partial response.
PFS | 1 year
  Progression-free survival.The time of patients from randomization to death caused by the progression of the tumor or any cause
OS | 3 year
  Overrall survival.The time of patient from randomization to death caused by any cause
QLQ | 3 year
  Quality of Life Questionnaire Core 30
the rate of incidence of adverse events | 3 year
  NCI CTC AE 4.03

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Medical University Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No